CLINICAL TRIAL: NCT05159219
Title: A Vanguard, Double-blind, Randomized, Placebo-controlled, Phase 2 Pilot Study to Investigate Prevention of Cardiovascular Events with Oral Colchicine 0.5mg Once Daily Compared with Placebo in Participants with Spontaneous ICH and Established, or Risk Factors For, Atherosclerosis
Brief Title: Colchicine for the Prevention of Vascular Events After an Acute Intracerebral Hemorrhage
Acronym: CoVasc-ICH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CoVasc-ICH
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial Hemorrhage; Colchicine
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Feasibility, double-blind, placebo-controlled randomized controlled trial (RCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product, with matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Colchicine, 0.5mg once daily (Experimental): Active colchicine tablet
  Interventions: Drug: Colchicine Pill
- Oral matching placebo, once daily (Placebo Comparator): Matching placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colchicine Pill — Anti-inflammatory
  Arms: Oral Colchicine, 0.5mg once daily
Other: Placebo — Inert ingredients
  Arms: Oral matching placebo, once daily

SUMMARY:
The overall goal is to establish the safety and efficacy of colchicine in ICH patients for the prevention of major cardiovascular events and brain injury. Colchicine for the prevention of vascular events after an acute intracerebral hemorrhage (CoVasc-ICH) is a vanguard pilot trial designed to obtain the factual feasibility prerequisites essential for the planning, design, funding and execution of a subsequent phase III trial.

ELIGIBILITY:
Inclusion Criteria

Adult participants are eligible to be included in the study only if all of the following criteria apply:

Type of Participant and Disease Characteristics

1. Participants with documented spontaneous intraparenchymal hemorrhage within 48 hours of symptom onset (or last seen normal) and
2. Qualifying for at least one of the following categories:

   i. history of symptomatic coronary, peripheral and/or carotid artery disease (severe atherosclerotic vascular disease), or ii. visualized extracranial cervical/intracranial atherosclerotic disease causing any degree of stenosis/occlusion or presence of aortic arch plaque with maximum thickness ≥1 mm (moderate atherosclerotic vascular disease), or iii. two or more risk factors including: age 60 years or older, hypertension, dyslipidemia, diabetes mellitus, chronic kidney disease (eGFR: 15-50mL/min), history of ischemic stroke or current smoking (mild atherosclerotic vascular disease)

   Informed Consent
3. Capable of giving signed informed consent either independently, or by a legally authorized representative (LAR), which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Secondary causes of ICH (relating to trauma, macrovascular anomalies, neoplasms or bleeding diathesis)
2. Inflammatory bowel disease or chronic diarrhea
3. Cirrhosis or severe hepatic dysfunction
4. Renal insufficiency (eGFR <15mL/min)

   Prior/Concomitant Therapy
5. Concurrent treatment with strong CYP3A4 inhibitors (atazanavir, clarithromycin, darunavir/ritonavir, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, tipranavir/ritonavir) or P-gp inhibitors (cyclosporine, ranolazine)
6. Known allergy or sensitivity to colchicine
7. Strong indication for colchicine where assignment to placebo is deemed unacceptable

   Other Exclusions
8. Pregnant or breast-feeding
9. Inability to adhere to study procedures
10. Estimated life expectancy less than 6 months at the time of enrollment
11. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g., employee or student of the investigational site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | From site activation until the end of recruitment (approximately 18 months)
  Recruitment Rate, mean of approximately 10 participants per site, per year

SECONDARY OUTCOMES:
Feasibility - Refusal Rate | Exploratory, from first patient, first visit, until the common study end date (approximately 30 months)
  Refusal to participate is not a substantial barrier to recruitment
Feasibility - Retention Rate | At 6 months from randomization
  Retention of ≥90% of study participants
Feasibility - Medication Adherence | At 12 months from randomization
  Adherence >75%

CONTACTS AND LOCATIONS:
Overall Officials: Aristeidis Katsanos, MD, Principal Investigator — Population Health Research Institute; Ashkan Shoamanesh, MD, Principal Investigator — Population Health Research Institute
Locations (11):
- Canada (11):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston Health Sciences, Kingston, Ontario
  - London Health Science Centre, University Hospital, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - University of Montreal, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilkinson CM, Katsanos AH, Sander NH, Kung TFC, Colbourne F, Shoamanesh A. Colchicine pre-treatment and post-treatment does not worsen bleeding or functional outcome after collagenase-induced intracerebral hemorrhage. PLoS One. 2022 Oct 18;17(10):e0276405. doi: 10.1371/journal.pone.0276405. eCollection 2022. PMID 36256671